CLINICAL TRIAL: NCT05326399
Title: Renal Biopsies in Post-liver Transplantation Patients With Renal Impairment: a Single-center, Prospective Cohort Study
Brief Title: Renal Biopsies in Post-liver Transplantation Patients With Renal Impairment
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shan Mou, Professor, RenJi Hospital
Other Study IDs: Renji20220326
Record Dates: First submitted 2022-03-26; First posted 2022-04-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Liver Transplantation; Renal Insufficiency, Chronic
Keywords: Liver transplantation; renal biopsy; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum and urine for laboratory examination
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- renal biopsy: Standard percutaneous biopsy has been performed in all participants. Light microscope, fluorescence microscope and electron microscope were used for assessment of kidney issue
  Interventions: Behavioral: renal biospy

INTERVENTIONS:
Behavioral: renal biospy — Standard percutaneous biopsy has been performed in all participants. Modification of treatment will be jointly decided by hepatologists and nephrologists based on the pathological results. All participants will be followed up for 96 weeks.

SUMMARY:
Investigators will conduct this single-center, prospective cohort study to explore the prevalence and risk factors of renal function progression in post-liver transplantation patients with renal impairment after renal biospy and to understand the the pathology of kidney disease in post-liver transplantation patients with renal impairment.

DETAILED DESCRIPTION:
This is a single-center, prospective, cohort study. This study will include approximate 369 post-liver transplantation patients with renal impairment and have received renal biopsy. Demographic characteristics, medical history, etiology of liver failure, concomitant medications, baseline laboratory parameters, etc., will be recorded. All participants will receive standard treatment by hepatologists and nephrologists based on the pathological results. All participants will be followed up for 96 weeks. Renal function, concomitant medications, and other laboratory parameters, etc., will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* patients received liver transplantation
* new onset of proteinuria(defined as 24-hour proteinuria>1g/24h, or Urinary albumin creatinine ratio(UACR)>300mg/g on at least two occasions), and/or renal impairment: eGFR <60 mL/min/1.73 m² at least two occasions, and/or serum creatinine increase ≥50% from baseline
* have received renal biopsy in the past 3 months
* Signed informed consent form(ICF)

Exclusion Criteria:

* patients received renal transplantation
* hepatic failure
* severe bleeding risk or platelet <70*109/L
* chronic kidney insufficiency with eGFR<30ml/min·1.73m2,or kidney atrophy, or solitary kidney, or medullary sponge kidney, or polycystic kidney, or obstructive nephropathy
* uncontrolled mental disease or unable to cooperate during operation
* Pregnancy or lactation
* not suitable for this study judged by investigaters

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients received liver transplantation with renal function and received renal biopsy
Sampling Method: Non-Probability Sample
Enrollment: 369 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression of renal function | 96 weeks
  Describe the cumulative incidence of renal function progression in post-liver transplantation patients with renal impairment after renal biopsy. Renal function progression is defined as a composite of end-starge renal disease(ESRD) or >100% increase of serum creatinine(Scr) or >50% per year decline of estimated glomerular filtration rate (eGFR)

SECONDARY OUTCOMES:
Risk factors of renal function deterioration in post-liver transplantation with renal impairment after renal biopsy | 96 weeks
  Investigate the risk factors of renal function deterioration in post-liver transplantation patients with renal impairment after renal biospy. Renal function deterioration is defined as a composite of ESRD or >100% increase of Scr or >50% per year decline of eGFR.
Pathology of kidney disease | 96 weeks
  Describe the pathology of kidney disease in post-liver transplantation patients with renal impairment.
Patient survival in post-liver transplantation patients with renal impairment after renal biopsy | 96 weeks
  Describe the patient survival rate in post-liver transplantation patients with renal impairment after renal biopsy.
Kidney survival in post-liver transplantation patients with renal impairment after renal biopsy | 96 weeks
  Describe the kidney survival rate in post-liver transplantation patients with renal impairment.
Remission of renal disease in post-liver transplantation patients with renal impairment after renal bisopy. | 96 weeks
  To describe the remission rate of renal disease in post-liver transplantation patients with renal impairment after renal biopsy. Remission is defined as 24-hour proteinuria decrease to <0.3g/24h or <50%of baseline, with stable kidney function(eGFR decrease less than 15%)
Effect of acute liver failure before liver trasplatation on renal impairment | 96 weeks
  Investigate the effect of acute liver failure before liver trasplatation on renal impairment with subgroup analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ojo AO, Held PJ, Port FK, Wolfe RA, Leichtman AB, Young EW, Arndorfer J, Christensen L, Merion RM. Chronic renal failure after transplantation of a nonrenal organ. N Engl J Med. 2003 Sep 4;349(10):931-40. doi: 10.1056/NEJMoa021744. PMID 12954741
- [Background] Neau-Cransac M, Morel D, Bernard PH, Merville P, Revel P, Potaux L, Saric J. Renal failure after liver transplantation: outcome after calcineurin inhibitor withdrawal. Clin Transplant. 2002 Oct;16(5):368-73. doi: 10.1034/j.1399-0012.2002.02028.x. PMID 12225434
- [Background] Welker MW, Weiler N, Bechstein WO, Herrmann E, Betz C, Schoffauer M, Zeuzem S, Sarrazin C, Amann K, Jung O. Key role of renal biopsy in management of progressive chronic kidney disease in liver graft recipients. J Nephrol. 2019 Feb;32(1):129-137. doi: 10.1007/s40620-018-0506-2. Epub 2018 Jun 26. PMID 29946864
- [Background] Chan GS, Lam MF, Kwan L, Fung SH, Chan SC, Chan KW. Clinicopathological study of renal biopsies after liver transplantation. Hong Kong Med J. 2013 Feb;19(1):27-32. PMID 23378351
- [Background] Lee JH, Cho YH, Ryu SJ, Kim SS, Lee YH, Jang IA, Choi BS, Choi JY, Kim DG, Choi YJ, Yang CW, Chung BH. Clinical usefulness of kidney biopsy in liver transplant recipients with renal impairment. Kidney Res Clin Pract. 2013 Dec;32(4):153-7. doi: 10.1016/j.krcp.2013.08.002. Epub 2013 Oct 24. PMID 26877934
- [Background] Kim JY, Akalin E, Dikman S, Gagliardi R, Schiano T, Bromberg J, Murphy B, de Boccardo G. The variable pathology of kidney disease after liver transplantation. Transplantation. 2010 Jan 27;89(2):215-21. doi: 10.1097/TP.0b013e3181c353e5. PMID 20098285
- [Background] O'Riordan A, Dutt N, Cairns H, Rela M, O'Grady JG, Heaton N, Hendry BM. Renal biopsy in liver transplant recipients. Nephrol Dial Transplant. 2009 Jul;24(7):2276-82. doi: 10.1093/ndt/gfp112. Epub 2009 Mar 16. PMID 19293134
- [Background] Bennett WM. Insights into chronic cyclosporine nephrotoxicity. Int J Clin Pharmacol Ther. 1996 Nov;34(11):515-9. PMID 8937936
- [Background] Pillebout E, Nochy D, Hill G, Conti F, Antoine C, Calmus Y, Glotz D. Renal histopathological lesions after orthotopic liver transplantation (OLT). Am J Transplant. 2005 May;5(5):1120-9. doi: 10.1111/j.1600-6143.2005.00852.x. PMID 15816895
- [Background] Fujinaga K, Usui M, Yamamoto N, Ishikawa E, Nakatani A, Kishiwada M, Mizuno S, Sakurai H, Tabata M, Isaji S. Hypertension and hepatitis C virus infection are strong risk factors for developing late renal dysfunction after living donor liver transplantation: significance of renal biopsy. Transplant Proc. 2014 Apr;46(3):804-10. doi: 10.1016/j.transproceed.2013.11.103. PMID 24767353
- [Background] Pichler RH, Huskey J, Kowalewska J, Moiz A, Perkins J, Davis CL, Leca N. Kidney Biopsies May Help Predict Renal Function After Liver Transplantation. Transplantation. 2016 Oct;100(10):2122-8. doi: 10.1097/TP.0000000000001334. PMID 27479161